CLINICAL TRIAL: NCT02082535
Title: S100B as a Marker of Brain Injury of Preterm Infants
Acronym: PTS100B
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Omer Bar-Yosef, Physician, Sheba Medical Center
Other Study IDs: SHEBA-13-0044-0B-CTIL
Record Dates: First submitted 2014-02-11; First posted 2014-03-10 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Premature Birth; Brain Injuries; Leukomalacia Periventricular; Developmental Disabilities
Keywords: Premature Birth; Brain Injuries; Leukomalacia Periventricular; S100B protein human; Glial Fibrillary Acidic Protein; Magnetic Resonance Imaging; Developmental Disabilities
MeSH Terms: conditions — Premature Birth; Brain Injuries; Leukomalacia, Periventricular; Developmental Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The improvement of treatment of preterm neonates improved their survival, however there is still significant portion of preterm infants (specifically very preterm infants) that suffers from brain insults and as a result developmental deficits. The brain injury is a consequence of hypoxic ischemic events, intracranial hemorrhages, as well as, infections and metabolic crisis. The brain injury is a combination of abnormal myelination, axonal damage and neuronal death. Although there is reduction in focal brain injury, diffuse brain injury is still abundant. Several treatments has been suggested and tested in animal models to prevent the brain insults including glutamate receptor blockers, allopurinol, xenon and different types of stem cells. However, two main obstacles prevent the use of these medication, first the uncertainty of their effect on the developing brain and second the difficulty to time the brain insult. Unlike neonatal asphyxia, when the delivery time and clinical signs are used to time and grade the brain injury, in preterm infants there is no real time tool to indicate severity and timing of brain injury. The disability point out a beneficial therapeutic window is a major obstacle in the acute treatment of brain injury in preterm infants. The aim of this study is to try and delineate such therapeutic window by using brain injury biomarkers.

S100b and GFAP are well recognized biomarkers of brain injury in adults, children and infants. Serial measurements of S100b in saliva (every 2 days) and GFAP in serum (weekly) will be sampled. A database of the clinical status of the infants will be collected, as well as, head ultra sound weekly and head MRI a term age. Development will be assessed by at 18 months. Two hypotheses are stated: One, increase in the levels of S100b and GFAP in their timing will be correlated with the severity of the clinical status, Two the duration of increased level of S100b and GFAP will be associated with abnormal MRI at term findings and abnormal developmental assessment.

ELIGIBILITY:
Inclusion Criteria:

- Preterm delivery before 30 week gestational age

Exclusion Criteria:

* Dysmorphic features in initial neurological examination
* Antenatal brain injury on fetal MRI or ultrasound
* Brain malformation
* Maternal drug abuse
* Maternal use of teratogenic medications

Ages: 1 Day to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Very early preterm infants born before 30 weeks gestational age
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
MRI at term age | 2-3 month after recruitment
  MRI description according to the protocol suggested by woodward et. al. (2006)
S100b and GFAP | 2-3 months after recruitment
  The level of S100b in a sample of 0.5 cc saliva will collected every 2 days and GFAP every week from the day of birth to discharge

SECONDARY OUTCOMES:
Developmental assessment at 18 month | 21 month after recruitment
  Neurological examination Griffith mental developmental scales (GMD-2) Vineland adaptive behavioral scale (VinelandTM-II) Clinical Adaptive Test/Clinical Linguistic and Auditory Milestone Scale
Developmental assessment at 3 month corrected age | 5-6 months after recuitment
  Neurological examination General Movements assessment Griffith mental developmental scales (GMD-2) Clinical Adaptive Test/Clinical Linguistic and Auditory Milestone Scale

CONTACTS AND LOCATIONS:
Overall Officials: Omer Bar Yosef, M.D. Ph.D., Principal Investigator — Sheba Medical Center, Ramat Gan, Israel
Locations (1):
- Sheba medical center, Ramat Gan, Israel